CLINICAL TRIAL: NCT03571802
Title: The Need of Dosing Adjustment for Simvastatin in Obese Patients Post Bariatric Surgery- Laparoscopic Sleeve Gastrectomy (LSG)
Brief Title: Pharmacokinetics of Simvastatin Post Laparoscopic Sleeve Gastrectomy (LSG)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSGSIMVASTATIN
Record Dates: First submitted 2018-05-22; First posted 2018-06-28 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Obesity; Hyperlipidemias
Keywords: pharmacokinetics; simvastatin; bariatric surgery; laparoscopic sleeve gastrectomy
MeSH Terms: conditions — Obesity; Hyperlipidemias | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic parameters of simvastatin before and after laparoscopic sleeve gastrectomy will be compared in 10 patients. Each patient will serve as their own control for comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- intervention arm (Experimental): simvastatin 20mg once
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — * The subject will take simvastatin 20mg at 0 h (after stopping simvastatin for 5 days). 5 mL of blood will be sampled at 0 h, 1 h, 2 h, 3 h, 5 h, 7 h.
  * There will be 2 blood sampling sessions: 1 before and the other 3 months after surgery.
  Other Names: Study arm

SUMMARY:
This study aims to investigate the change in systemic exposure of simvastatin post LSG.

DETAILED DESCRIPTION:
Morbid obesity (Body mass index > 40 kg/m2 or 35-39 kg/m2 with comorbidity; 37.5 kg/m2 for Asians) is a growing global health issue. Bariatric surgery is the only intervention that has demonstrated sustainable reduction in weight and comorbidities.1,2 Among the various bariatric procedures, laparoscopic sleeve gastrectomy (LSG) has rapidly gained popularity worldwide.3,4 Physiological alterations following LSG include reduction in gastrointestinal surface and reduced retention of food. Bioavailability of drugs may be affected but published literature in this area is sparse and studies are usually small and uncontrolled.5-7 Moreover, some reports concerning gastric banding and jejunoileal bypass are no longer practiced because of the associated risk. In general, bioavailability of orally administered drug changes with a reduction in gastrointestinal area. While Kroll et al showed slight increase in area under curve of rivaroxaban post bariatric surgery8, Skottheim et al demonstrated significant but variable change in systemic exposure of atorvastatin after gastric bypass (from threefold decrease to twofold increase) that diminished but was sustained with time (21-45 months post gastric bypass)9-10.

No study has investigated the change in pharmacokinetics of simvastatin post LSG.

Simvastatin is a widely-used lipid-lowering agent with a low bioavailability of 5% due to the extensive first pass metabolism.11 As simvastatin undergoes hydrolysis in the stomach to the active form12, it is postulated that bioavailability of simvastatin will decrease after LSG.13-15 A decrease in bioavailability may be associated with reduced efficacy. Authors of review articles suggested choosing an alternative agent to simvastatin post bariatric surgery. However, such recommendation is largely based on theoretical concern rather than solid evidence.14,15 A previous study attempted to model the pharmacokinetics of simvastatin post Roux-en-Y and biliopancreatic diversion with duodenal switch.13 The data is not applicable to LSG and the model did not take into account of the pH-dependent hydrolysis. This will be the first study aiming to investigate the change in systemic exposure of simvastatin post LSG.

ELIGIBILITY:
Inclusion Criteria:

* Planned for laparoscopic sleeve gastrectomy at National University Hospital
* Taking statin
* Aged 21 or above

Exclusion Criteria:

* Patient on concomitant treatment with medications/ food/ herbal supplements that may affect the pharmacokinetics of simvastatin: boceprevir, conivaptan, cyclosporine, efavirenz, mitotane, tocilizumab, rifamycin, amiodarone, amlodipine, aprepitant, azithromycin, colchicine, fenofibrate, imatinib, raltegravir, ranolazine, teriflunomide, ticagrelor, fusidic acid, protease inhibitors, telaprevir, telithromycin, gemfibrozil, erythromycin, clarithromycin, carbamazepine, rifampicin, ketoconazole, fluconazole, itraconazole, voriconanzole, diltiazem, verapamil, dexamethasone, prednisolone, phenytoin, ritonavir, indinavir, nelfinavir, bosentan, telithromycin, nefazodone, St John's wort, orlistat, sibutramine and other strong CYP 3A4 inhibitors/ inducers
* Pregnant ladies

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of simvastatin | baseline (before surgery). 3 months after surgery
  Ratio of AUC of simvastatin for each subject before and 3 months after surgery will be calculated, the mean ratio will be reported
Maximum serum concentration (Cmax) of simvastatin | baseline (before surgery). 3 months after surgery
  Ratio of Cmax of simvastatin for each subject before and 3 months after surgery will be calculated, the mean ratio will be reported
Time at which maximum serum concentration (Tmax) of simvastatin | baseline (before surgery). 3 months after surgery
  Ratio of Tmax of simvastatin for each subject before and 3 months after surgery will be calculated, the mean ratio will be reported
Area Under Curve (AUC) of simvastatin acid | baseline (before surgery). 3 months after surgery
  Ratio of AUC of simvastatin acid for each subject before and 3 months after surgery will be calculated, the mean ratio will be reported
Maximum serum concentration (Cmax) of simvastatin acid | baseline (before surgery). 3 months after surgery
  Ratio of Cmax of simvastatin acid for each subject before and 3 months after surgery will be calculated, the mean ratio will be reported
Time at which maximum serum concentration (Tmax) of simvastatin acid | baseline (before surgery). 3 months after surgery
  Ratio of Tmax of simvastatin acid for each subject before and 3 months after surgery will be calculated, the mean ratio will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Asim Shabbir, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Skottheim IB, Stormark K, Christensen H, Jakobsen GS, Hjelmesaeth J, Jenssen T, Reubsaet JL, Sandbu R, Asberg A. Significantly altered systemic exposure to atorvastatin acid following gastric bypass surgery in morbidly obese patients. Clin Pharmacol Ther. 2009 Sep;86(3):311-8. doi: 10.1038/clpt.2009.82. Epub 2009 Jun 3. PMID 19494810
- [Background] Jakobsen GS, Skottheim IB, Sandbu R, Christensen H, Roislien J, Asberg A, Hjelmesaeth J. Long-term effects of gastric bypass and duodenal switch on systemic exposure of atorvastatin. Surg Endosc. 2013 Jun;27(6):2094-101. doi: 10.1007/s00464-012-2716-3. Epub 2012 Dec 18. PMID 23247745

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT03571802/Prot_SAP_000.pdf